CLINICAL TRIAL: NCT07285824
Title: Virtual McKenzie Exercises and Centralization of Pain: A Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Evidence In Motion (Other)
Collaborators: University of Nevada, Las Vegas (Other); College of St. Scholastica, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VirtualMcKenzie2025
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain; Low Back Pain
Keywords: Low Back Pain; Chronic Pain; Directional Preference; McKenzie Method; Extension-Based Exercise; Motor Imagery; Virtual Exercise; Pain Centralization; Fear-Avoidance; Pain Catastrophization; Physical Therapy; Cortical Representation; Somatosensory Cortex (S1); Body Schema; Disability
MeSH Terms: conditions — Chronic Pain; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motor Imagery Extension Protocol (Experimental): Participants with low back pain who demonstrate a directional preference for extension will receive a single session of a guided motor imagery protocol simulating lumbar extension movements based on the McKenzie method. The intervention is designed to mentally replicate an extension press-up without requiring physical movement.
  Interventions: Behavioral: Motor Imagery-Based Lumbar Extension

INTERVENTIONS:
Behavioral: Motor Imagery-Based Lumbar Extension — Participants will lie prone with hands positioned under the shoulders in a standard "pre-press-up" position. With eyes closed, participants will be verbally guided through ten imagined lumbar extension press-ups. The standardized motor imagery script includes:
  Focusing attention on current back and leg symptoms
  Imagining pushing the arms into extension
  Visualizing the back arching into extension
  Holding the imagined end-range position for several seconds
  Imagining returning to the starting position in a controlled manner
  Repeating this process ten times
  Total duration of the protocol is approximately 5 minutes.
  Mode of Delivery:
  In-person, guided by a physical therapist trained in the study protocol.
  Purpose:
  To evaluate immediate changes in pain, disability, psychological measures, physical mobility, neurodynamic measures, and symptom centralization following a motor imagery-based extension intervention.

SUMMARY:
Low back pain (LBP) is frequently managed in physical therapy using the McKenzie method, in which a patient's directional preference-most commonly extension-is used to guide treatment. Extension-based interventions are associated with symptom improvement and centralization in many individuals with LBP. At the same time, research in pain neuroscience has shown that people with LBP may have altered cortical representations of the low back, which may contribute to pain and disability. For patients who experience high pain levels or significant fear of movement, active directional preference exercises may be difficult to perform.

Motor imagery, the mental simulation of movement without physical execution, has been shown to activate brain regions involved in movement and may help modify altered cortical representations. Preliminary research has suggested that virtual or imagery-based McKenzie extension exercises may improve pain and movement-related outcomes.

This exploratory study aims to evaluate the immediate effects of a brief motor imagery-based extension protocol in adults with LBP who demonstrate a directional preference for extension. The study will assess changes in pain intensity, disability, fear-avoidance, pain catastrophization, lumbar flexion, straight leg raise, pain distribution, and symptom centralization following a single motor imagery session.

DETAILED DESCRIPTION:
Background and Rationale:

Low back pain (LBP) is the most common musculoskeletal condition treated in outpatient physical therapy, accounting for approximately 25-40% of patient visits. Directional preference, a key element of the McKenzie method, is widely used in the management of LBP. This approach assesses how a patient's symptoms respond to repeated or sustained directional movements-most commonly flexion or extension-and integrates the direction that reduces or centralizes symptoms into the treatment plan. Previous research demonstrates that extension-based directional preference strategies are effective for a large proportion of patients with LBP and are associated with pain reduction, increased mobility, reduced fear of movement, and centralization of radiating symptoms.

In parallel with traditional mechanical assessment and treatment methods, pain neuroscience research has highlighted the role of changes in cortical body maps, particularly in the primary somatosensory cortex (S1), in individuals with LBP. People with persistent LBP exhibit altered S1 representations, including changes in size and organization of cortical maps, which are associated with pain, disability, and functional limitations. These representations are dynamic, and movement-based therapies can help normalize them.

However, patients with high pain levels, significant fear-avoidance, or sensitized nervous systems may find movement-based interventions difficult to perform. Motor imagery-mentally simulating movement without performing it physically-may provide an alternative method for modifying cortical representations while reducing threat and avoiding symptom aggravation. Motor imagery activates neural regions similar to those used during actual movement execution and may be beneficial for individuals reluctant to engage in active movement.

Preliminary findings have suggested that virtual or imagery-based McKenzie extension movements may improve pain, fear-avoidance, catastrophization, and mobility in individuals with LBP. Because centralization of symptoms is a hallmark feature of directional preference-based care, this study aims to further explore whether a brief motor imagery-based extension protocol can influence pain intensity, body pain distribution, psychological constructs, physical measures, and centralization in patients with LBP who demonstrate an extension directional preference.

Study Objectives:

The primary objective of this study is to evaluate the immediate effects of a guided motor imagery extension protocol in patients with LBP who demonstrate a directional preference for extension. The study aims to determine whether the intervention results in changes in pain intensity, disability, fear-avoidance, pain catastrophization, lumbar flexion, straight leg raise, and pain distribution, as well as whether patients report centralization of symptoms.

Study Design:

This study is a single-group, pre-post exploratory design conducted across three outpatient physical therapy clinics. Institutional Review Board approval will be obtained prior to study initiation. Eligible patients presenting with LBP will be identified during their initial evaluation. Participants must be between 18 and 65 years of age, able to read and understand English, present with no red flags during review of systems, have no prior spinal surgery, and demonstrate a positive response to extension-based directional preference testing. Participation is voluntary and requires written informed consent.

Intervention Procedures:

Following consent, participants will complete a demographics questionnaire. A blinded therapist will administer baseline measures including disability, pain intensity, fear-avoidance beliefs, pain catastrophization, active trunk flexion, straight leg raise (SLR), and a pain body chart.

Participants will then receive a brief educational explanation of cortical map changes associated with LBP. Next, participants will assume a prone "pre-press-up" position, placing their hands under their shoulders. Instead of performing an active press-up, they will close their eyes and receive verbal guidance through a series of ten motor imagery-based lumbar extension movements. The standardized script instructs participants to visualize completing a full press-up, experiencing spinal extension, holding briefly at end range, and returning to the starting position. Total intervention time is approximately five minutes.

Immediately following the imagery protocol, a blinded therapist will repeat all outcome measures. After data collection, clinicians will resume their usual plan of care for each patient.

Outcome Measures:

Pre- and post-intervention measures include:

Oswestry Disability Index (ODI) to assess functional disability

Numeric Pain Rating Scale (NPRS) for low back and leg pain

Fear Avoidance Beliefs Questionnaire (FABQ), including Physical Activity and Work subscales

Pain Catastrophization Scale (PCS)

Active lumbar flexion (fingertip-to-floor distance in centimeters)

Straight Leg Raise measured with an inclinometer

Body chart with grid overlay to quantify pain distribution and potential changes in cortical representation

Data Management and Analysis:

De-identified data will be compiled and analyzed using descriptive statistics for demographic variables. Pre- and post-intervention comparisons will be performed using paired-samples t-tests with significance set at p < 0.05. Significant findings will be confirmed with Wilcoxon Signed Ranks nonparametric testing.

ELIGIBILITY:
Inclusion Criteria:

Age 18 to 65 years

Presenting to outpatient physical therapy with low back pain (LBP)

Able to read and understand English

No red flags identified during review of systems and initial physical therapy evaluation

No prior spinal surgery

Demonstrates a positive response to extension-based directional preference testing

Willing and able to provide written informed consent

Exclusion Criteria:

Age younger than 18 or older than 65

Inability to read or understand English

Presence of red flags during review of systems (e.g., suspected fracture, malignancy, infection, cauda equina symptoms)

History of spinal surgery

No demonstrable directional preference for extension during evaluation

Any condition that the evaluating clinician determines would preclude safe participation

Declines to participate or is unable to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Low Back Pain Intensity (NPRS - Low Back) | Pre-intervention to immediately post-intervention (same session).
  Change in self-reported low back pain intensity measured using the 0-10 Numeric Pain Rating Scale (NPRS), where 0 = no pain and 10 = worst imaginable pain.
Leg Pain Intensity (NPRS - Leg) | Pre-intervention to immediately post-intervention (same session).
  Change in self-reported leg pain intensity using the 0-10 NPRS.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Pre-intervention to immediately post-intervention.
  Change in disability level measured by the 10-item ODI questionnaire. Scores range from 0-50, multiplied by 2 to produce a percentage (0-100%), with higher scores indicating greater disability.
Fear-Avoidance Beliefs Questionnaire (FABQ) - Physical Activity Subscale | Pre-intervention to immediately post-intervention.
  Change in fear-avoidance beliefs related to work. The 7-item FABQ-W yields scores from 0-42, with higher scores indicating greater work-related fear-avoidance.
Pain Catastrophization Scale (PCS) | Pre-intervention to immediately post-intervention.
  Change in pain catastrophizing as measured by the 13-item PCS. Total scores range from 0-52, with higher scores indicating greater catastrophic thinking about pain.
Active Lumbar Flexion (Fingertip-to-Floor Distance) | Pre-intervention to immediately post-intervention.
  Change in active trunk forward flexion measured in centimeters from the tip of the longest finger of the dominant hand to the floor. Lower values indicate greater lumbar and hamstring mobility.
Straight Leg Raise (SLR) | Pre-intervention to immediately post-intervention.
  Change in SLR measured using an inclinometer placed on the tibia. SLR is measured on the most affected leg, with the ankle maintained in neutral. Degrees of hip flexion are recorded.
Pain Distribution (Body Chart Grid Count) | Pre-intervention to immediately post-intervention.
  Change in pain distribution measured using a standardized body chart. Pain areas are quantified using a grid overlay, producing a count of regions marked by the participant.
Symptom Centralization (Qualitative Report) | Immediately post-intervention.
  Presence or absence of centralization of symptoms based on patient self-report during or after the motor imagery extension protocol. Centralization is defined as a proximal shift of pain toward the lumbar spine.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerhardt A, Eich W, Janke S, Leisner S, Treede RD, Tesarz J. Chronic Widespread Back Pain is Distinct From Chronic Local Back Pain: Evidence From Quantitative Sensory Testing, Pain Drawings, and Psychometrics. Clin J Pain. 2016 Jul;32(7):568-79. doi: 10.1097/AJP.0000000000000300. PMID 26379077
- [Background] Sanders NW, Mann NH 3rd, Spengler DM. Pain drawing scoring is not improved by inclusion of patient-reported pain sensation. Spine (Phila Pa 1976). 2006 Nov 1;31(23):2735-41; discussion 2742-3. doi: 10.1097/01.brs.0000244674.99258.f9. PMID 17077744
- [Background] Lacey RJ, Lewis M, Jordan K, Jinks C, Sim J. Interrater reliability of scoring of pain drawings in a self-report health survey. Spine (Phila Pa 1976). 2005 Aug 15;30(16):E455-8. doi: 10.1097/01.brs.0000174274.38485.ee. PMID 16103839
- [Background] Matthews M, Rathleff MS, Vicenzino B, Boudreau SA. Capturing patient-reported area of knee pain: a concurrent validity study using digital technology in patients with patellofemoral pain. PeerJ. 2018 Mar 8;6:e4406. doi: 10.7717/peerj.4406. eCollection 2018. PMID 29568700
- [Background] Wand BM, Keeves J, Bourgoin C, George PJ, Smith AJ, O'Connell NE, Moseley GL. Mislocalization of sensory information in people with chronic low back pain: a preliminary investigation. Clin J Pain. 2013 Aug;29(8):737-43. doi: 10.1097/AJP.0b013e318274b320. PMID 23835768
- [Background] Ekedahl H, Jonsson B, Frobell RB. Fingertip-to-floor test and straight leg raising test: validity, responsiveness, and predictive value in patients with acute/subacute low back pain. Arch Phys Med Rehabil. 2012 Dec;93(12):2210-5. doi: 10.1016/j.apmr.2012.04.020. Epub 2012 Apr 30. PMID 22555005
- [Background] Zimney K, Louw A, Puentedura EJ. Use of Therapeutic Neuroscience Education to address psychosocial factors associated with acute low back pain: a case report. Physiother Theory Pract. 2014 Apr;30(3):202-9. doi: 10.3109/09593985.2013.856508. Epub 2013 Nov 19. PMID 24252071
- [Background] George SZ, Valencia C, Beneciuk JM. A psychometric investigation of fear-avoidance model measures in patients with chronic low back pain. J Orthop Sports Phys Ther. 2010 Apr;40(4):197-205. doi: 10.2519/jospt.2010.3298. PMID 20357418
- [Background] Moseley GL. Evidence for a direct relationship between cognitive and physical change during an education intervention in people with chronic low back pain. Eur J Pain. 2004 Feb;8(1):39-45. doi: 10.1016/S1090-3801(03)00063-6. PMID 14690673
- [Background] Moseley GL, Nicholas MK, Hodges PW. A randomized controlled trial of intensive neurophysiology education in chronic low back pain. Clin J Pain. 2004 Sep-Oct;20(5):324-30. doi: 10.1097/00002508-200409000-00007. PMID 15322439
- [Background] Burton AK, Waddell G, Tillotson KM, Summerton N. Information and advice to patients with back pain can have a positive effect. A randomized controlled trial of a novel educational booklet in primary care. Spine (Phila Pa 1976). 1999 Dec 1;24(23):2484-91. doi: 10.1097/00007632-199912010-00010. PMID 10626311
- [Background] Fritz JM, George SZ. Identifying psychosocial variables in patients with acute work-related low back pain: the importance of fear-avoidance beliefs. Phys Ther. 2002 Oct;82(10):973-83. PMID 12350212
- [Background] Poiraudeau S, Rannou F, Baron G, Henanff LA, Coudeyre E, Rozenberg S, Huas D, Martineau C, Jolivet-Landreau I, Garcia-Mace J, Revel M, Ravaud P. Fear-avoidance beliefs about back pain in patients with subacute low back pain. Pain. 2006 Oct;124(3):305-311. doi: 10.1016/j.pain.2006.04.019. Epub 2006 Jun 5. PMID 16740362
- [Background] Grotle M, Vollestad NK, Brox JI. Clinical course and impact of fear-avoidance beliefs in low back pain: prospective cohort study of acute and chronic low back pain: II. Spine (Phila Pa 1976). 2006 Apr 20;31(9):1038-46. doi: 10.1097/01.brs.0000214878.01709.0e. PMID 16641782
- [Background] Cleland JA, Fritz JM, Childs JD. Psychometric properties of the Fear-Avoidance Beliefs Questionnaire and Tampa Scale of Kinesiophobia in patients with neck pain. Am J Phys Med Rehabil. 2008 Feb;87(2):109-17. doi: 10.1097/PHM.0b013e31815b61f1. PMID 17993982
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Cleland JA, Childs JD, Whitman JM. Psychometric properties of the Neck Disability Index and Numeric Pain Rating Scale in patients with mechanical neck pain. Arch Phys Med Rehabil. 2008 Jan;89(1):69-74. doi: 10.1016/j.apmr.2007.08.126. PMID 18164333
- [Background] Moseley GL. Widespread brain activity during an abdominal task markedly reduced after pain physiology education: fMRI evaluation of a single patient with chronic low back pain. Aust J Physiother. 2005;51(1):49-52. doi: 10.1016/s0004-9514(05)70053-2. PMID 15748125
- [Background] Moseley L. Combined physiotherapy and education is efficacious for chronic low back pain. Aust J Physiother. 2002;48(4):297-302. doi: 10.1016/s0004-9514(14)60169-0. PMID 12443524
- [Background] Hakkinen A, Kautiainen H, Jarvenpaa S, Arkela-Kautiainen M, Ylinen J. Changes in the total Oswestry Index and its ten items in females and males pre- and post-surgery for lumbar disc herniation: a 1-year follow-up. Eur Spine J. 2007 Mar;16(3):347-52. doi: 10.1007/s00586-006-0187-8. Epub 2006 Aug 16. PMID 16912888
- [Background] Fritz JM, Irrgang JJ. A comparison of a modified Oswestry Low Back Pain Disability Questionnaire and the Quebec Back Pain Disability Scale. Phys Ther. 2001 Feb;81(2):776-88. doi: 10.1093/ptj/81.2.776. PMID 11175676
- [Background] Deyo RA, Battie M, Beurskens AJ, Bombardier C, Croft P, Koes B, Malmivaara A, Roland M, Von Korff M, Waddell G. Outcome measures for low back pain research. A proposal for standardized use. Spine (Phila Pa 1976). 1998 Sep 15;23(18):2003-13. doi: 10.1097/00007632-199809150-00018. PMID 9779535
- [Background] Louw A, Farrell K, Landers M, Barclay M, Goodman E, Gillund J, McCaffrey S, Timmerman L. The effect of manual therapy and neuroplasticity education on chronic low back pain: a randomized clinical trial. J Man Manip Ther. 2017 Dec;25(5):227-234. doi: 10.1080/10669817.2016.1231860. Epub 2016 Sep 22. PMID 29449764
- [Background] Louw A, Goldrick S, Bernstetter A, Van Gelder LH, Parr A, Zimney K, Cox T. Evaluation is treatment for low back pain. J Man Manip Ther. 2021 Feb;29(1):4-13. doi: 10.1080/10669817.2020.1730056. Epub 2020 Feb 24. PMID 32091317
- [Background] Louw A, Farrell K, Nielsen A, O'Malley M, Cox T, Puentedura EJ. Virtual McKenzie extension exercises for low back and leg pain: a prospective pilot exploratory case series. J Man Manip Ther. 2023 Feb;31(1):46-52. doi: 10.1080/10669817.2022.2092822. Epub 2022 Jun 23. PMID 35739614
- [Background] Gallese V, Fadiga L, Fogassi L, Rizzolatti G. Action recognition in the premotor cortex. Brain. 1996 Apr;119 ( Pt 2):593-609. doi: 10.1093/brain/119.2.593. PMID 8800951
- [Background] Lotze M, Halsband U. Motor imagery. J Physiol Paris. 2006 Jun;99(4-6):386-95. doi: 10.1016/j.jphysparis.2006.03.012. Epub 2006 May 22. PMID 16716573
- [Background] Moseley GL. Graded motor imagery is effective for long-standing complex regional pain syndrome: a randomised controlled trial. Pain. 2004 Mar;108(1-2):192-8. doi: 10.1016/j.pain.2004.01.006. PMID 15109523
- [Background] Vlaeyen JW, Crombez G. Fear of movement/(re)injury, avoidance and pain disability in chronic low back pain patients. Man Ther. 1999 Nov;4(4):187-95. doi: 10.1054/math.1999.0199. PMID 10593107
- [Background] Vlaeyen JWS, Kole-Snijders AMJ, Boeren RGB, van Eek H. Fear of movement/(re)injury in chronic low back pain and its relation to behavioral performance. Pain. 1995 Sep;62(3):363-372. doi: 10.1016/0304-3959(94)00279-N. PMID 8657437
- [Background] Lloyd D, Findlay G, Roberts N, Nurmikko T. Differences in low back pain behavior are reflected in the cerebral response to tactile stimulation of the lower back. Spine (Phila Pa 1976). 2008 May 20;33(12):1372-7. doi: 10.1097/BRS.0b013e3181734a8a. PMID 18496351
- [Background] Flor H, Elbert T, Muhlnickel W, Pantev C, Wienbruch C, Taub E. Cortical reorganization and phantom phenomena in congenital and traumatic upper-extremity amputees. Exp Brain Res. 1998 Mar;119(2):205-12. doi: 10.1007/s002210050334. PMID 9535570
- [Background] Moseley GL. Distorted body image in complex regional pain syndrome. Neurology. 2005 Sep 13;65(5):773. doi: 10.1212/01.wnl.0000174515.07205.11. No abstract available. PMID 16157921
- [Background] Lotze M, Moseley GL. Role of distorted body image in pain. Curr Rheumatol Rep. 2007 Dec;9(6):488-96. doi: 10.1007/s11926-007-0079-x. PMID 18177603
- [Background] Moseley LG. I can't find it! Distorted body image and tactile dysfunction in patients with chronic back pain. Pain. 2008 Nov 15;140(1):239-243. doi: 10.1016/j.pain.2008.08.001. Epub 2008 Sep 10. PMID 18786763
- [Background] Maihofner C, Neundorfer B, Birklein F, Handwerker HO. Mislocalization of tactile stimulation in patients with complex regional pain syndrome. J Neurol. 2006 Jun;253(6):772-9. doi: 10.1007/s00415-006-0117-z. Epub 2006 May 18. PMID 16705476
- [Background] Flor H, Braun C, Elbert T, Birbaumer N. Extensive reorganization of primary somatosensory cortex in chronic back pain patients. Neurosci Lett. 1997 Mar 7;224(1):5-8. doi: 10.1016/s0304-3940(97)13441-3. PMID 9132689
- [Background] Holmes NP, Spence C. The body schema and the multisensory representation(s) of peripersonal space. Cogn Process. 2004 Jun;5(2):94-105. doi: 10.1007/s10339-004-0013-3. PMID 16467906
- [Background] Stavrinou ML, Della Penna S, Pizzella V, Torquati K, Cianflone F, Franciotti R, Bezerianos A, Romani GL, Rossini PM. Temporal dynamics of plastic changes in human primary somatosensory cortex after finger webbing. Cereb Cortex. 2007 Sep;17(9):2134-42. doi: 10.1093/cercor/bhl120. Epub 2006 Nov 16. PMID 17110591
- [Background] Flor H. The functional organization of the brain in chronic pain. Prog Brain Res. 2000;129:313-22. doi: 10.1016/S0079-6123(00)29023-7. No abstract available. PMID 11098699
- [Background] Wand BM, Parkitny L, O'Connell NE, Luomajoki H, McAuley JH, Thacker M, Moseley GL. Cortical changes in chronic low back pain: current state of the art and implications for clinical practice. Man Ther. 2011 Feb;16(1):15-20. doi: 10.1016/j.math.2010.06.008. Epub 2010 Jul 23. PMID 20655796
- [Background] Nijs J, Roussel N, Paul van Wilgen C, Koke A, Smeets R. Thinking beyond muscles and joints: therapists' and patients' attitudes and beliefs regarding chronic musculoskeletal pain are key to applying effective treatment. Man Ther. 2013 Apr;18(2):96-102. doi: 10.1016/j.math.2012.11.001. Epub 2012 Dec 28. PMID 23273516
- [Background] Donelson R, Aprill C, Medcalf R, Grant W. A prospective study of centralization of lumbar and referred pain. A predictor of symptomatic discs and anular competence. Spine (Phila Pa 1976). 1997 May 15;22(10):1115-22. doi: 10.1097/00007632-199705150-00011. PMID 9160470
- [Background] Namnaqani FI, Mashabi AS, Yaseen KM, Alshehri MA. The effectiveness of McKenzie method compared to manual therapy for treating chronic low back pain: a systematic review. J Musculoskelet Neuronal Interact. 2019 Dec 1;19(4):492-499. PMID 31789300
- [Background] Karlsson M, Bergenheim A, Larsson MEH, Nordeman L, van Tulder M, Bernhardsson S. Effects of exercise therapy in patients with acute low back pain: a systematic review of systematic reviews. Syst Rev. 2020 Aug 14;9(1):182. doi: 10.1186/s13643-020-01412-8. PMID 32795336
- [Background] Surkitt LD, Ford JJ, Hahne AJ, Pizzari T, McMeeken JM. Efficacy of directional preference management for low back pain: a systematic review. Phys Ther. 2012 May;92(5):652-65. doi: 10.2522/ptj.20100251. Epub 2012 Jan 12. PMID 22247407
- [Background] May S, Aina A. Centralization and directional preference: a systematic review. Man Ther. 2012 Dec;17(6):497-506. doi: 10.1016/j.math.2012.05.003. Epub 2012 Jun 12. PMID 22695365
- [Background] Kuhnow A, Kuhnow J, Ham D, Rosedale R. The McKenzie Method and its association with psychosocial outcomes in low back pain: a systematic review. Physiother Theory Pract. 2021 Dec;37(12):1283-1297. doi: 10.1080/09593985.2019.1710881. Epub 2020 Jan 7. PMID 31910720
- [Background] Nechvatal P, Hitrik T, Kendrova LD, Macej M. Comparison of the effect of the McKenzie method and spiral stabilization in patients with low back pain: A prospective, randomized clinical trial. J Back Musculoskelet Rehabil. 2022;35(3):641-647. doi: 10.3233/BMR-210055. PMID 34657873
- [Background] Long A, Donelson R, Fung T. Does it matter which exercise? A randomized control trial of exercise for low back pain. Spine (Phila Pa 1976). 2004 Dec 1;29(23):2593-602. doi: 10.1097/01.brs.0000146464.23007.2a. PMID 15564907
- [Background] May S, Rosedale R. An international survey of the comprehensiveness of the McKenzie classification system and the proportions of classifications and directional preferences in patients with spinal pain. Musculoskelet Sci Pract. 2019 Feb;39:10-15. doi: 10.1016/j.msksp.2018.06.006. Epub 2018 Jun 19. PMID 30447492
- [Background] Halliday MH, Pappas E, Hancock MJ, Clare HA, Pinto RZ, Robertson G, Ferreira PH. A Randomized Controlled Trial Comparing the McKenzie Method to Motor Control Exercises in People With Chronic Low Back Pain and a Directional Preference. J Orthop Sports Phys Ther. 2016 Jul;46(7):514-22. doi: 10.2519/jospt.2016.6379. Epub 2016 May 12. PMID 27170524
- [Background] Hefford C. McKenzie classification of mechanical spinal pain: profile of syndromes and directions of preference. Man Ther. 2008 Feb;13(1):75-81. doi: 10.1016/j.math.2006.08.005. Epub 2006 Dec 22. PMID 17188547
- [Background] George SZ, Fritz JM, Silfies SP, Schneider MJ, Beneciuk JM, Lentz TA, Gilliam JR, Hendren S, Norman KS. Interventions for the Management of Acute and Chronic Low Back Pain: Revision 2021. J Orthop Sports Phys Ther. 2021 Nov;51(11):CPG1-CPG60. doi: 10.2519/jospt.2021.0304. PMID 34719942
- [Background] Zheng P, Kao MC, Karayannis NV, Smuck M. Stagnant Physical Therapy Referral Rates Alongside Rising Opioid Prescription Rates in Patients With Low Back Pain in the United States 1997-2010. Spine (Phila Pa 1976). 2017 May 1;42(9):670-674. doi: 10.1097/BRS.0000000000001875. PMID 28441685